CLINICAL TRIAL: NCT00551642
Title: The Effects of Nitric Oxide for Inhalation on the Development of Chronic Lung Disease in Pre-term Infants
Brief Title: Safety and Efficacy Study of Nitric Oxide for Inhalation on Chronic Lung Disease in Premature Babies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INOT27; 2004-002312-29 (EudraCT Number)
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Results first posted 2010-10-18 (Estimated); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Lung Disease
Keywords: Preemie, Inhaled Nitric Oxide
MeSH Terms: conditions — Lung Diseases | interventions — Nitric Oxide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhaled Nitric Oxide (INO) (Active Comparator): INO administered by nasal continuous positive airway pressure, nasal cannula or face mask at 5 parts per million (ppm) for between 7 and 21 days
  Interventions: Drug: Nitric oxide
- Placebo (Placebo Comparator): Placebo gas administered by nasal continuous positive airway pressure, nasal cannula or face mask, for a maximum of 21 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitric oxide — Nitric Oxide vapour (gas) for inhalation (400 ppm)
  Other Names: INO max®
  Arms: Inhaled Nitric Oxide (INO)
Drug: Placebo — Placebo gas for inhalation
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of inhaled nitric oxide to reduce the risk of chronic lung disease in pre-term infants with respiratory distress, and to assess the long-term effects of the therapy on the development of these children over 7 years of clinical follow-up.

DETAILED DESCRIPTION:
Although the effects of inhaled Nitric Oxide on pulmonary vascular tone are well-described and relevant to term infants with persistent pulmonary hypertension, the pathophysiology of respiratory failure in preterm infants may be quite different. Chronic lung disease (CLD) represents the final pathway of a heterogeneous group of pulmonary disorders of infancy that usually start in the neonatal period. CLD most commonly occurs in preterm (<30 weeks of gestational age (GA) infants with birth weights less than 1,500 grams (g), and especially in those very preterm (<26 weeks GA) with birth weights less than 1,000 g, and who have been treated for respiratory distress syndrome (RDS).

ELIGIBILITY:
Inclusion Criteria:

* Inborn preterm infants 24+0 weeks-28+6 days weeks gestational age (defined by first trimester ultrasound or if not available based on the last menstrual period) who requires the use of surfactant within 24 hours of birth (either prophylactically, or for signs of developing respiratory distress), or who requires the use of continuous positive airway pressure (CPAP) (fraction of inspired oxygen concentration (FiO2) ≥ 0.30 on a mean airway pressure ≥ 4cm water (H2O)) within 24 hours of birth in order to maintain an oxygen saturation (SpO2) ≥ 85%.
* Informed consent of the guardian.

Exclusion Criteria:

* Outborn infants.
* Infants ≥ 29 weeks gestational age.
* Infants requiring FiO2 >0.5 to maintain SpO2 >85%, on a sufficient mean airway pressure (e.g., > 8 cm H2O on controlled mechanical ventilation (CMV)) in order to achieve adequate chest inflation (8-9 ribs on Chest X-ray) two hours after the proper administration of exogenous surfactant.
* Any suspected congenital heart disease other than patent ductus arteriosus or atrial septal defect.
* Any infant with severe bleeding or coagulation abnormalities at high-risk of diathesis, e.g., platelet <50,000 per millimeter cube (mm³), fibrinogen <0.5 gram per liter (g/L), other clotting factors <10%.
* Any infant in whom a decision has been made not to provide full treatment, e.g., chromosomal abnormalities, severe multiple abnormalities, severe birth asphyxia, etc.
* Use of another investigational drug or device before or during the active study period.

Max Age: 26 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 800 (Actual)
Dates: Start 2005-05-29 (Actual); Primary Completion 2008-03-16 (Actual); Study Completion 2015-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Director — Mallinckrodt
Locations (35):
- Belgium (4):
  - UCL St. LUC, Brussels
  - Clinique Notre Dame, Charleroi
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Clinique St. Vincent CHC, Rocourt
- Oulun yliopsistollinen sairaala, Oulu, Finland
- France (3):
  - Centre Hospitalier Intercommunal de Creteil, Créteil
  - Hospital Mere-Enfant, Nantes
  - Hospital Robert Debre, Paris
- Germany (7):
  - Campus Charite Mitte, Berlin
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Mannheim, Mannheim
  - Universitaetsklinikum Marburg, Marburg
  - Universitaetsklinikum Muenchen, München
  - Universitaeklinikum Tuebingen, Tübingen
  - Univeritaetsklinik Ulm, Ulm
- Italy (6):
  - Az. Osp. G. Salesi, Ancona
  - Ospedali Riuniti, Bergamo
  - Policlinico S. Orsola, Bologna
  - Azienda Ospedaliera Careggi, Florence
  - University Padova, Padua
  - Policlinico Gemelli, Roma
- Netherlands (2):
  - Beatrix Children's Hospital, University Medical Center Groningen, Groningen
  - Sophia Kinderziekenhuis, Rotterdam
- Spain (7):
  - Hospital de Cruces, Barakaldo
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Gregorio Mar, Madrid
  - Hosspital Univeritario La Paz, Madrid
  - Hospital Universitario Canarias, Santa Cruz de Tenerife
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario La Fe, Valencia
- Sweden (2):
  - Astrid Lindgrens barnsjukjus, Karolinska Unviersritets sjukhuset-Solna, Stockholm
  - Akademiska Sjukhuset, Uppsala
- United Kingdom (3):
  - Meedway Mariton Hospital, Gillingham
  - Leicester Royal Infirmary, Leicester
  - Kings College, London

IPD SHARING:
Plan to Share IPD: No
Discussion of statistical endpoints and analysis are included in manuscripts. Summary aggregate (basic) results (including adverse events information) and the study protocol are made available on clinicaltrials.gov (NCT00551642) when required by regulation. Individual de-identified patient data will not be disclosed. Requests for additional information should be directed to the company at medinfo@mnk.com.

REFERENCES:
- [Derived] Laube M, Amann E, Uhlig U, Yang Y, Fuchs HW, Zemlin M, Mercier JC, Maier RF, Hummler HD, Uhlig S, Thome UH. Inflammatory Mediators in Tracheal Aspirates of Preterm Infants Participating in a Randomized Trial of Inhaled Nitric Oxide. PLoS One. 2017 Jan 3;12(1):e0169352. doi: 10.1371/journal.pone.0169352. eCollection 2017. PMID 28046032
- [Derived] Durrmeyer X, Hummler H, Sanchez-Luna M, Carnielli VP, Field D, Greenough A, Van Overmeire B, Jonsson B, Hallman M, Mercier JC, Marlow N, Johnson S, Baldassarre J; European Union Nitric Oxide Study Group. Two-year outcomes of a randomized controlled trial of inhaled nitric oxide in premature infants. Pediatrics. 2013 Sep;132(3):e695-703. doi: 10.1542/peds.2013-0007. Epub 2013 Aug 12. PMID 23940237
- [Derived] Mercier JC, Hummler H, Durrmeyer X, Sanchez-Luna M, Carnielli V, Field D, Greenough A, Van Overmeire B, Jonsson B, Hallman M, Baldassarre J; EUNO Study Group. Inhaled nitric oxide for prevention of bronchopulmonary dysplasia in premature babies (EUNO): a randomised controlled trial. Lancet. 2010 Jul 31;376(9738):346-54. doi: 10.1016/S0140-6736(10)60664-2. Epub 2010 Jul 23. PMID 20655106

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-five Medical Centers participated and enrolled a total of 800 participants (Intent to treat population).
Pre-assignment Details: 800 participants were enrolled at 35 medical centers around the world for the Treatment period, and 305 had data at the 7-year Follow-up period.
Groups:
- Inhaled Nitric Oxide (INO): INO administered by nasal continuous positive airway pressure, nasal cannula or face mask at 5 parts per million (ppm) for between 7 and 21 days during the Treatment period, but no intervention during the 7-year Follow-up
- Placebo: Placebo gas administered by nasal continuous positive airway pressure, nasal cannula or face mask, for a maximum of 21 days during the Treatment period, but no intervention during the 7-year Follow-up
Period: Treatment Period
Arm/Group | Inhaled Nitric Oxide (INO) | Placebo
Started | 399 | 401
Safety Population | 395 | 397
Completed | 338 | 338
Not Completed | 61 | 63
Not completed — Protocol Deviation | 6 | 11
Not completed — Delivery device failure | 1 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Death | 33 | 31
Not completed — Inclusion/Exclusion criteria | 4 | 4
Not completed — Adverse Event | 15 | 12
Not completed — Withdrawal by Subject | 2 | 1
Period: 7-Year Follow-up
Arm/Group | Inhaled Nitric Oxide (INO) | Placebo
Started (Participants with data available at 7-year Follow-up) | 152 | 153
Completed | 152 | 153
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Nitric Oxide (INO) | Placebo | Total
Number analyzed (Participants) | 399 | 401 | 800
Age, Customized [Count of Participants; unit: Participants]
  Preterm newborn infants (gestational age < 37 wks) | 399 | 401 | 800
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 192 | 181 | 373
  Male | 207 | 220 | 427

OUTCOME MEASURES:

1. Primary Outcome: Survival Without Bronchopulmonary Dysplasia (BPD) in Preterm Infants With Respiratory Distress
Description: Survival without BPD is defined as the number of preterm infants of 36 weeks gestational age who survived the treatment period without the need for supplemental oxygen
Time Frame: 21 days
Population: All participants with efficacy data
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (INO) | Placebo
Number analyzed (Participants) | 395 | 400
Participants | 258 | 262
Statistical Analysis 1: Comparison: Inhaled Nitric Oxide (INO) vs Placebo; Test type: Other; p = 0.7340, Wald Chi-square; Odds Ratio (OR) = 1.05

2. Other Pre Specified Outcome: Mortality at 7-year Follow-up
Description: Number of participants who died between 2 years and the 7-year Follow-up Period
Time Frame: at 7-year Follow-up
Population: Participants with 7-year follow-up data
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (INO) | Placebo
Number analyzed (Participants) | 152 | 153
Participants | 0 | 0

3. Other Pre Specified Outcome: Strengths and Difficulties Questionnaire Results for Participants at 7-year Follow-up
Description: The Strengths and Difficulties Questionnaire contained 25 questions that were used to create 5 scales (ranging from 10=most normal to 0=most abnormal) for emotional symptoms, conduct problems, hyperactivity, peer problems, and (10=most abnormal, 0=most normal) for prosocial.
Time Frame: At 7-year Follow-up
Population: Participants with Questionnaire Results at the 7-year follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inhaled Nitric Oxide (INO) | Placebo
Number analyzed (Participants) | 147 | 147
score on a scale
  Emotional (0=most normal, 10=most abnormal) | 1.9 (1.79) | 2.1 (1.96)
  Conduct (0=most normal, 10=most abnormal) | 1.4 (1.55) | 1.4 (1.58)
  Hyperactivity (0=most normal, 10=most abnormal) | 3.8 (2.64) | 3.4 (2.66)
  Peer problems (0=most normal, 10=most abnormal) | 1.2 (1.41) | 1.5 (1.74)
  Prosocial (10=most abnormal, 0=most normal) | 8.6 (1.73) | 8.4 (1.81)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs), including clinically significant changes in vital signs, oxygen saturation, and laboratory values, were collected in the safety population for a maximum of 21 days (not during follow-up). All serious AEs are listed, and non-serious treatment-emergent adverse events (TEAEs) are listed if 5% or more participants in any arm experienced any form of that preferred term within 21 days. Survival was counted through the 7-year follow-up, and included under All-cause Mortality.
Description: In a previous submission of this record, "Survival", "Vital Signs", "Arterial Oxygen Saturation by Pulse Oximetry", "Adverse Events" and "Methemoglobin Level" were incorrectly included as Outcome Measures, but have been deleted from the current version, because clinically significant changes in these parameters were counted under adverse events and/or all-cause mortality presented in this adverse events module.
Groups:
- Placebo: Placebo gas administered by nasal continuous positive airway pressure (nasal cannula or face mask) for a maximum of 21 days during the Treatment period, but no intervention during the 7-year Follow-up
Arm/Group | Inhaled Nitric Oxide (INO) | Placebo
All-Cause Mortality (participants affected / at risk) | 56/395 | 48/397
Serious Adverse Events (participants affected / at risk) | 170/395 | 177/397
Other Adverse Events (participants affected / at risk) | 358/395 | 334/397
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Nitric Oxide (INO) (N=395) | Placebo (N=397)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest neonatal (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Coarctation of the aorta (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 62 (62) | 54 (54)
Persistent foetal circulation (Congenital, familial and genetic disorders) | 2 (2) | 0 (0)
Vitello-intestinal duct remnant (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 1 (1)
Retinopathy of prematurity (Eye disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal perforation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (2)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 17 (17) | 14 (14)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0)
Meconium ileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Meconium plug syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 16 (16) | 9 (9)
Oesophageal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 1 (1)
Volvulus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Catheter related complication (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Gallbladder perforation (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 34 (35) | 35 (39)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Feeding tube complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bacterial test positive (Investigations) | 1 (1) | 0 (0)
Blood cortisol decreased (Investigations) | 0 (0) | 1 (1)
Blood growth hormone decreased (Investigations) | 0 (0) | 1 (1)
Brain scan abnormal (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hepatic haemangioma rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Central nervous system lesion (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ventricle dilatation (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 50 (52) | 42 (42)
Hydrocephalus (Nervous system disorders) | 4 (4) | 4 (4)
Periventricular leukomalacia (Nervous system disorders) | 7 (7) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 4 (4)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Foreign body aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 13 (15)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 14 (14)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Pulmonary interstitial emphysema syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chest tube insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 4 (4) | 1 (1)
Infarction (Vascular disorders) | 1 (1) | 2 (2)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Nitric Oxide (INO) (N=395) | Placebo (N=397)
Anaemia (Blood and lymphatic system disorders) | 189 (253) | 168 (226)
Thrombocytopenia (Blood and lymphatic system disorders) | 29 (29) | 28 (31)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 183 (187) | 158 (163)
Hyperbilirubinaemia (Hepatobiliary disorders) | 122 (138) | 120 (130)
Jaundice (Hepatobiliary disorders) | 98 (107) | 89 (97)
Sepsis (Infections and infestations) | 68 (75) | 60 (66)
Hyperglycaemia (Metabolism and nutrition disorders) | 90 (100) | 68 (75)
Hyponatraemia (Metabolism and nutrition disorders) | 21 (22) | 19 (21)
Metabolic acidosis (Metabolism and nutrition disorders) | 49 (53) | 52 (62)
Haemorrhage intracranial (Nervous system disorders) | 73 (81) | 55 (58)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 73 (78) | 78 (79)
Hypotension (Vascular disorders) | 55 (57) | 50 (54)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other